CLINICAL TRIAL: NCT00875238
Title: Predicting Adverse Cardiac Events in Breast Cancer Therapy (PACE in Breast Cancer)
Brief Title: Side Effects Involving the Heart in Women With Breast Cancer Receiving Doxorubicin and Trastuzumab
Acronym: PACE in BC
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: CDR0000613213; P30CA068485 (NIH); VU-VICC-BRE-0767
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer; Cardiac Toxicity; Cardiovascular Complications
Keywords: cardiac toxicity; cardiovascular complications; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — Trastuzumab; Doxorubicin; Amplified Fragment Length Polymorphism Analysis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Mononuclear Cells
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: doxorubicin hydrochloride
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: magnetic resonance imaging

SUMMARY:
RATIONALE: Studying samples of blood and tissue in the laboratory from women receiving doxorubicin and trastuzumab for breast cancer may help doctors learn more about changes that occur in DNA and identify biomarkers for increased risk of cardiac effects.

PURPOSE: This clinical trial is studying side effects involving the heart in women with breast cancer receiving doxorubicin and trastuzumab.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if polymorphisms in genes (e.g., CYBA, RAC2, NCF4, MRP1, MRP2, GTSP and CBR3) in women with breast cancer treated with doxorubicin hydrochloride increase the relative risk of developing ≥ NCI grade 1 cardiotoxicity. (Primary study)
* To determine whether pre-treatment levels of biomarkers (e.g., neuregulin, IGF-1, cardiotrophin-1, IL-6, VEGF, hepatocyte growth factor, and heparin binding EGF) in these patients, correlate with relative risk of developing ≥ NCI grade 1 cardiotoxicity to this regimen. (Primary study)
* To determine whether decreased heart rate variability and increased plasma levels of norepinephrine at 3 weeks after completion of this regimen correlate with relative risk of developing ≥ NCI grade 1 cardiotoxicity in these patients. (Primary study)
* To determine whether decrease in endothelial progenitor cell (EPC) number at 3 weeks after completion of this regimen can be detected, and if so whether decreased EPC number correlates with ≥ NCI grade 1 cardiotoxicity. (Primary study)
* To determine whether baseline physical fitness level of these patients, assessed by a questionnaire and 6 minute walk distance, correlates with relative risk of developing ≥ NCI grade 1 cardiotoxicity to this regimen. (Primary study)
* To determine whether activity level of these patients during treatment, assessed by questionnaire, correlates with relative risk of developing ≥ NCI grade 1 cardiotoxicity to this regimen. (Primary study)
* To determine whether drop in functional capacity of these patients, measured by 6 minute walk distance at the end of treatment with this regimen, correlates with ≥ NCI grade 1 cardiotoxicity. (Primary study)
* To determine whether MRI can detect changes in diastolic heart function in these patients 48 hours after administration of this regimen. (Sub-study A)
* To determine if a greater decrease in diastolic dysfunction in these patients at 48 hours is predictive of greater decrease in systolic function at 3 weeks after treatment with this regimen. (Sub-study A)
* To determine whether levels of certain biomarkers of cardiac myocyte damage, B-type natriuretic peptide and the sarcomere protein troponin T at 48 hours after the initial exposure to these drugs correlate with relative risk of developing ≥ NCI grade1 cardiotoxicity. (Sub-study A)
* To determine whether trastuzumab given concurrently with doxorubicin hydrochloride decreases heart rate variability and increases plasma levels of norepinephrine in these patients, and if so, whether these changes correlate with relative risk of developing NCI grade ≥ 1 cardiotoxicity. (Sub-study B)
* To determine whether EPC number obtained from patients treated with trastuzumab have decreased migration into microvascular structures in an ex vivo assay and whether these changes correlate with ≥ NCI grade 1 cardiotoxicity. (Sub-study B)
* To determine whether levels of certain biomarkers in these patients , including neuregulin, IGF-1, cardiotrophin-1, IL-6, VEGF, hepatocyte growth factor and heparin binding EGF, change after exposure to trastuzumab. (Sub-study B)

OUTLINE: This is a multicenter study.

* Primary study: Patients make an initial visit (before beginning doxorubicin hydrochloride treatment) and a visit 3 weeks after the 4th course of doxorubicin hydrochloride (approximately 12 weeks after the initial visit). During these visits, blood samples are also collected for measuring serum levels of neuregulin-1, IGF-1, cardiotropin-1, IL-6, VEGF, hepatocyte growth factor, and plasma norepinephrine and endothelial progenitor cells (EPC). Heart-rate variability (HRV) is measured and, if necessary, a transthoracic echocardiogram is performed. Patients complete baseline health and activity level questionnaire and suitable patients complete a 6-minute walk test. Patients undergo blood collection for genotype analysis for single nucleotide polymorphism sites during the initial visit.

Patients complete a questionnaire assessing physical activity at the beginning of the 2nd, 3rd, and 4th courses of chemotherapy.

* Sub-study A (MRI)*: In addition to the assessments performed in the primary study, patients undergo some extra tests. During initial visit, patients have an additional blood sample collected during initial visit for measurement of B-type natriuretic peptide (BNP) and troponin T and undergo cardiac MRI. Approximately 48 hours after the first dose of doxorubicin hydrochloride, patients undergo an additional visit, during which blood samples are collected for BNP and troponin T and an cardiac MRI is performed.

NOTE: *Patients who enroll in sub-study A must also be enrolled in the primary study.

* Sub-study B (trastuzumab)*: In addition to the assessments performed in the primary study, patients undergo some extra tests. Patients undergo an additional visit after the third treatment of trastuzumab (approximately 6 months after the first dose of doxorubicin hydrochloride), during which patients have blood samples collected and analyzed as in Primary study visit 2. HRV is measured and, if necessary, a transthoracic echocardiogram is performed.

NOTE: *Patients who enroll in sub-study B must also be enrolled in the primary study.

After completion of study treatment, patients are followed periodically for up to 5 years .

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with breast cancer

  * Receiving treatment at Vanderbilt Ingram Cancer Center and other participating oncology practices in middle Tennessee and southern Kentucky
* Starting a standard doxorubicin hydrochloride regimen for 4 courses

  * Also scheduled to receive trastuzumab (for patients enrolled in sub-study B only)
* No presence of metastatic disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Karnofsky performance status 60-100%
* Not pregnant
* Negative pregnancy test
* Additional criteria for sub-study A (MRI):

  * Glomerular filtration rate ≥ 60 mL/min
  * No implanted electronic devices, cochlear implants, metallic implants, shrapnel or neurosurgical clips
  * No prior adverse reaction to gadolinium-based contrast agents
  * Must not exceed the weight limit or be too large to fit in the MRI scanner

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior anthracycline chemotherapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with newly diagnosed breast cancer with planned anthracycline-based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2008-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in cardiac function by echocardiogram | 5 years
  change in cardiac function as measured by serial echocardiograms

SECONDARY OUTCOMES:
Overall feasibility | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Carrie G Lenneman, MD, MSCI, Principal Investigator — Vanderbilt-Ingram Cancer Center & Univ. of Louisville; Daniel Lenihan, MD, Principal Investigator — Vanderbilt University; Douglas B Sawyer, MD, PhD, Principal Investigator — Vanderbilt University
Locations (4):
- United States (4):
  - University of Louisville James Graham Brown Cancer Center, Louisville, Kentucky
  - Vanderbilt Heart One Hundred Oaks, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Geisberg CA, Abdallah WM, da Silva M, Silverstein C, Smith HM, Abramson V, Mayer I, Means-Powell J, Freehardt D, White B, Lenihan D, Sawyer DB. Circulating neuregulin during the transition from stage A to stage B/C heart failure in a breast cancer cohort. J Card Fail. 2013 Jan;19(1):10-5. doi: 10.1016/j.cardfail.2012.11.006. PMID 23273589
- [Derived] Lenneman CG, Abdallah WM, Smith HM, Abramson V, Mayer IA, Silverstein C, Silverstein C, Means-Powell J, Paranjape SY, Lenihan D, Sawyer DB, Raj SR. Sympathetic nervous system alterations with HER2+ antagonism: an early marker of cardiac dysfunction with breast cancer treatment? Ecancermedicalscience. 2014 Jul 17;8:446. doi: 10.3332/ecancer.2014.446. eCollection 2014. PMID 25114718